CLINICAL TRIAL: NCT01867879
Title: A Phase 1 Study to Evaluate the Cardiac Safety of Orally Administered TAS-102 in Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate the Cardiac Safety of TAS-102 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TPU-TAS-102-103; 2013-000650-21 (EudraCT Number)
Record Dates: First submitted 2013-05-24; First posted 2013-06-04 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors (Excluding Breast Cancer)
Keywords: Advanced solid tumors (excluding breast cancer) for which no standard therapy exists
MeSH Terms: interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-102 — 35 mg/m2/dose, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: TAS-102
Drug: Placebo — Placebo tablets, orally, single dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the cardiac safety of TAS-102 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, nonrandomized study to evaluate the cardiac safety of TAS-102 in patients with advanced solid tumors. The study is conducted in 2 phases: the cardiac safety evaluation phase to investigate cardiac repolarization and the cardiac safety profile (Cycle 1) and the extension phase to assess the safety profile and antitumor activity (subsequent cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has advanced solid tumors (excluding breast cancer) for which no standard therapy exists
3. Has received no more than 5 prior cancer therapies
4. ECOG performance status of 0 or 1
5. Is able to take medications orally
6. Corrected QT interval using Bazett's correction is no more than 450 msec on resting ECG
7. Has adequate organ function (bone marrow, kidney and liver)
8. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has had certain other recent treatment e.g. major surgery, extended field radiation, anticancer therapy, received investigational agent, within the specified time frames prior to study drug administration
2. Certain serious illnesses or medical condition(s)
3. Has a family history of unexplained sudden death or long QT syndrome
4. Has had a documented cardiovascular complication following a fluoropyrimidine-derived treatment
5. Is a patient for whom it is not technically possible to obtain quality ECG tracings
6. Is receiving a concomitant drug that is known to affect QT interval or to be arrhythmogenic
7. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
8. Known sensitivity to TAS-102 or its components
9. Is a pregnant or lactating female
10. Refuses to use an adequate means of contraception (including male patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
QTc interval | Days -2, -1, 1, and 12 of Cycle 1
  Predose (Day -2) to post-dose changes and absolute values in QTc interval after placebo (Day -1, Cycle 1), after a single dose of TAS-102 (Day 1, Cycle 1), and after multiple doses (Day 12, Cycle 1)

SECONDARY OUTCOMES:
Quantitative and Qualitative ECG parameters | Days -2, -1, 1, and 12 of Cycle 1
  Predose (Day -2) to postdose changes and absolute values in quantitative Holter ECG parameters (heart rate, RR, PR and QRS intervals) after placebo (Day -1, Cycle 1), after a single dose of TAS-102 (Day 1, Cycle 1), and after multiple doses (Day 12, Cycle 1). In addition, qualitative assessments of Holter ECG recordings will be performed.
Relationship between TAS-102 pharmacokinetics and its effect on cardiac repolarization | Days 1 and 12 of Cycle 1
  Pharmacokinetic samples are taken on Days 1 and 12 of Cycle 1. The relationship between plasma concentrations of TAS-102 and the change from baseline in QTc adjusted by placebo will be quantified using a linear mixed effect model approach.
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) will be used.
Tumor assessments using Response Evaluation Criteria in Solid Tumors (RECIST) | Every 8 weeks through Cycle 6 (ie, through 24 weeks). Thereafter, assessments will be performed at least every 12 weeks according to site standard of care, until at least one of the treatment discontinuation criteria is met.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Bendell JC, Patel MR, Yoshida K, Seraj J, Weaver R, Lemech C, Todaro TG, Pant S, Arkenau HT. Phase 1 study of cardiac safety of TAS-102 in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Jun;77(6):1275-83. doi: 10.1007/s00280-016-3031-9. Epub 2016 May 5. PMID 27151157